CLINICAL TRIAL: NCT01671228
Title: Development of a Patient Decision Aid (PtDA) to Facilitate Renal Patients Informed Decisions About Dialysis Treatments
Brief Title: Developing and Evaluating the Yorkshire Dialysis Decision Aid
Acronym: YoDDA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Kidney Cancer UK (Other); National Health Service, United Kingdom (Other Government); Baxter Healthcare Corporation (Industry); Foundation for Informed Medical Decision Making (Other)
Responsible Party: Principal Investigator, Hilary L Bekker, Senior Lecturer in Behavioural Sciences and Chartered Psychologist, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: V4_01_JUN_12; SP2/Choices/2012 (Other Grant/Funding Number: Kidney Research UK); 0171-1 (Other Grant/Funding Number: Foundation of Informed Decision Making research grant)
Record Dates: First submitted 2012-08-16; First posted 2012-08-23 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Kidney Failure
Keywords: dialysis; chronic kidney failure; informed choice; patient decision making; decision aid
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- decision aid (Experimental): The Yorkshire Dialysis Decision Aid (YoDDA). Delivered as a leaflet in clinic and a web resource outside the NHS.
  Interventions: Other: Decision Aid
- Decision Aid + values task (Experimental): The Yorkshire Dialysis Decision Aid (YoDDA) + values clarification questions. delivered as a leaflet in clinic and a web-based resource outside the NHS.
  Interventions: Other: Decision Aid; Other: Decision Aid + values task
- Decision Aid + patient stories (Experimental): The Yorkshire Dialysis Decision Aid (YoDDA) + patient stories. Delivered as an web-based resource outside the NHS.
  Interventions: Other: Decision Aid; Other: Decision aid + patient stories
- usual predialysis education (No Intervention): The consultations and information usually provided by the predialysis health professionals

INTERVENTIONS:
Other: Decision Aid — The Yorkshire Dialysis Decision Aid (YoDDA) resource in web and paper format
  Arms: Decision Aid + patient stories; Decision Aid + values task; decision aid
Other: Decision aid + patient stories — The Yorkshire dialysis decision aid (YoDDA) plus a set of narratives provided by patients on the treatment options (home and hospital haemodialysis; continuous ambulatory and automated peritoneal dialysis
  Arms: Decision Aid + patient stories
Other: Decision Aid + values task — The Yorkshire Dialysis decision aid (YoDDA) plus a set of questions to help patients explore what aspects of their life important to them about this decision (values clarification)
  Arms: Decision Aid + values task

SUMMARY:
The purpose of this research is to develop a patient decision aid in paper and web formats to help patients with chronic kidney disease make informed dialysis treatment decisions.

DETAILED DESCRIPTION:
This research will develop and evaluate a paper and web resource known as a decision-aid to help patients make informed decisions about dialysis treatment. The Yorkshire Dialysis Decision Aid (YoDDA) will help patients' with chronic kidney disease make informed decisions between haemodialysis and peritoneal dialysis choices by a) re-writing dialysis information in a more meaningful way for patients, b) restructuring information to make this difficult decision more manageable, and c) using prompts to help patients imagine the choices' consequences. The research will assess the acceptability of a patient decision aid in paper and web versions to patients and their carers, and its impact on patients choices about dialysis.

The programme of research included:

A survey using qualitative methods of patients with chronic kidney disease and professionals providing predialysis services to develop the Yorkshire Dialysis Decision Aid content, and integration within usual predialysis care practices.

A before-and-after study was carried out to evaluate the acceptability of the YoDDA-booklet to patients with sustained deterioration of kidney function making dialysis decision across the Yorkshire and Humber region, UK.

An experimental study was carried out on-line to evaluate the acceptability of three versions of YoDDA-web (YoDDA; YoDDA+values tasks; YoDDA_patient videos) to people, or carers of people, with kidney disease. The study was advertised with flyers within UK renal units and notices on the National Kidney Federation's website and members' magazine.

ELIGIBILITY:
Inclusion Criteria: Adult patients with chronic kidney disease and carers of people with chronic kidney diseae who are making decisions about dialysis treatments.

-

Exclusion Criteria: Those not literate in English

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2011-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Preparation for decision making scale | one and six weeks after provision information about dialysis choices
  Assesses patient's perception of how useful the resource was in helping patients prepare for a consultation to talk about their health decision (Graham and O'Connor, 2010). http://decisionaid.ohri.ca/docs/develop/User_Manuals/UM_PrepDM.pdf

SECONDARY OUTCOMES:
Usefulness of information | one and six weeks after the provision of information
  Study specific items to assess perceived usefulness of information in helping patients understand chronic kidney disease, dialysis treatments and thinking about dialysis

OTHER OUTCOMES:
Dialysis treatment preferences | one week and six weeks after the information
  Study specific measure asking patients to rank order their preferred dialysis treatment (CAPD, APD, home HD, centre HD)

CONTACTS AND LOCATIONS:
Overall Officials: Hilary L Bekker, PhD, Principal Investigator — University of Leeds
Locations (6):
- United Kingdom (6):
  - Hull and East Yorkshire Hospital Trust, Hull, East Yorkshire
  - Sheffield Northern General Teaching Hospital, Sheffield, South Yorkshire
  - St James University Hospital, Leeds, West Yorkshire
  - Bradford Teaching Hospital, Bradford, Yorkshire
  - York teaching Hospital NHS Foundation trust, York, Yorkshire
  - Doncaster Royal Infirmary, Doncaster